CLINICAL TRIAL: NCT05247541
Title: Diagnosing Chronic Exertional Compartment Syndrome: Measurement of Intra-Compartmental Pressures Using Noninvasive Subharmonic Aided Pressure Estimation (SHAPE) Versus Shear Wave Elastography (SWE).
Brief Title: Diagnosing Compartment Syndrome With SHAPE vs Elastography
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Lantheus Medical Imaging (Industry); Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Flemming Forsberg, Professor, Thomas Jefferson University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CG20003
Record Dates: First submitted 2022-01-27; First posted 2022-02-21 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Chronic Exertional Compartment Syndrome
MeSH Terms: conditions — Chronic Exertional Compartment Syndrome | interventions — perflutren

STUDY DESIGN:
Intervention Model Description: This study will be performed as a prospective nonblinded pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Participants (Active Comparator)
  Interventions: Drug: Definity
- Study participants (Experimental)
  Interventions: Drug: Definity

INTERVENTIONS:
Drug: Definity — Definity (Lantheus Medical Imaging, N Billerica, MA) in 50 mL of saline infused over 5-10 minutes

SUMMARY:
Chronic exertional compartment syndrome (CECS) is an innocuous condition seen primarily in 10-60% of young active people with exercise induced leg pain. With an average delay in diagnosis of 2 years, early identification is crucial as delays have led to poor surgical outcomes after fasciotomy. Diagnosis is currently made by compartment pressure (CP) testing, which is invasive, painful and demonstrates variable accuracy. There is no literature on the role of shear wave elastography (SWE) and/or subharmonic assisted pressure estimation (SHAPE) with microbubbles in diagnosing CECS. Ultrasound contrast agents are FDA-approved and are extremely safe. In this single-blinded prospective pilot study, the accuracy of SHAPE and SWE will be evaluated and compared to the current gold standard of compartment testing in patients with suspected CECS. Muscle stiffness and record a quantitative assessment of enhancement and hydrostatic pressures will be documented and correlated with compartment testing results based on a reference standard modified Pedowitz criteria for CECS

DETAILED DESCRIPTION:
Chronic exertional compartment syndrome (CECS) is an innocuous condition seen primarily in 10-60% of young, active people with exercise induced leg pain. Patients present with anterior lower extremity pain that worsens with exercise and resolves after rest. CECS arises from increased intra-compartmental pressure causing impaired tissue perfusion. The average delay in diagnosis and subsequent treatment is 2 years, which has been shown to decrease the success rate of both conservative and surgical therapy. Definitive treatment is with fasciotomy, which has a success rate of up to 95%.

The etiology of CECS is not well understood but is thought to arise from volume expansion of a muscle within a noncompliant space bounded by fascia and bone resulting in insufficient blood flow and a resultant oxygen supply and demand mismatch in that compartment. In some cases the physiological response may lead to a 20% increase in muscle volume. Several risk factors have been identified including pre- existing fascial defects (seen in 40% of CECS patients) and a smaller capillary density to muscle size ratio. In rare cases, CECS may progress to acute compartment syndrome - a surgical emergency requiring emergent fasciotomy.

The gold standard for diagnosing CECS is direct measurement of intra-compartmental pressures with maximum sensitivity and specificity in recent studies of 93% and 74%. However, in rare circumstances, diagnosis can be made on clinical basis alone. Compartment pressure testing is performed by inserting a handheld large gauge needle with a pressure monitor into the muscle and measuring the compartment pressure directly (in mmHg). Direct compartment testing is invasive, painful, and carries a complication risk of neurovascular damage and infection. Furthermore, there is significant variability in this technique with some studies finding more than >5 mmHg difference in 40% of compartmental pressure measurements.

In the diagnostic algorithm of CECS, imaging is primarily used to rule out other more common causes of lower extremity leg pain such as medial tibial stress syndrome (MTSS), stress fractures, and muscle strains. Several non-invasive imaging modalities have been used to diagnose CECS. When compared to pressure testing, MRI showed similar sensitivity, but lower specificity (< 60%). While MRI has shown some diagnostic promise, it is more expensive, less ubiquitous, and less accurate than compartment testing. Near-infrared spectroscopy, which measures hemoglobin O2 saturation of tissues, has shown to have clinically equivalent sensitivies (85%) compared to compartment testing, however, it is not readily available.

A clinical exam alone is insensitive and non-specific in the diagnosis of CECS. Therefore, surgeons must rely on a combination of clinical exam and imaging to determine whether a patient is a surgical candidate. An accurate, non-invasive, and cost effective diagnostic tool does not currently exist for patients with suspected CECS. SWE is a safe, non-invasive and relatively inexpensive modality that has wide ranging diagnostic capabilities. SWE is used measure liver stiffness thereby staging fibrosis in chronic liver disease, following up previously diagnosed hepatic fibrosis and evaluating patients with portal hypertension. Recently, the utility of SWE in musculoskeletal imaging has increased; for example SWE is currently being using to evaluate tendinopahic achilles tendons with some clinical success.

FDA-approved ultrasound contrast agents are safe, non-nephrotoxic, non-hepatotoxic contrast agents that act as echo-enhancers before dissipation from the intravascular space. SHAPE utilizing microbubbles has been used for the noninvasive estimation of hydrostatic blood pressure to monitor interstitial fluid pressure in tumors, assess the degree of portal hypertension, and to monitor neoadjuvant chemotherapy for breast cancer patients. However, no series studies exist characterizing SHAPE and SWE for the screening or diagnosis of CECS. This study will assess whether SHAPE and/or SWE can accurately detect increased intra-compartmental pressures when compared to the reference standard of intra-compartmental pressure testing.

This study will be performed as a prospective single-blinded pilot study of patients with suspected CECS who is eligible to participate in the study and meets inclusion and exclusion criteria (described below). A research Coordinator will meet with the patient to explain the study in full. If the prospective subject expresses interest in participating in the study an investigator will approach the patient to obtain consent. All sonographic research portions of the study will be performed by a certified and experienced sonographer. The compartment testing portion of the study will be performed as part of the subjects standard of care.

Pre-exercise SWE: After determining inclusion, patients will undergo pre-exercise SWE using a Logiq E10 ultrasound system (GE Healthcare, Waukesha WI) with a linear array transducer. All images will be obtained with the ankle in a neutral position. Conventional B-mode imaging will be used to identify the muscle of interest. Imaging will be used to guide placement of ROIs, which can be adjusted by the operator After shear waves have propagated through the muscle of concern tissue displacement maps are used to calculate shear-wave velocity in meters per second. Elasticity parameters, including mean (Emean), maximum (Emax), minimum (Emin), and standard deviation (ESD) will be displayed on the ultrasound machine monitor. Tissue stiffness will then be directly calculated, expressed as the shear modulus G in kilopascals (kPa). Quantitative shear modulus maps will be generated.

Pre-exercise SHAPE: The modified software allowing the E10 to operate in subharmonic imaging (SHI) mode will permit acquisition of subharmonic data. All images will be obtained with the ankle in the neutral position. An 18-24 gauge intravenous line will be placed in either the right or left Upper extremity. The contrast will be an intravenous infusion of 2 vials of Definity (Lantheus Medical Imaging, N Billerica, MA) in 50 mL of saline infused over 5-10 minutes. The route of administration and dosages follow the recommendations issued by the manufacturer. SHI will be performed using the same scanner. A broad bandwidth C2-9 convex probe will be used to acquire conventional and subharmonic images (transmitting at 5.8 MHz receiving at 2.9 MHz). The investigators will run a power optimization algorithm to establish individual acoustic parameters settings for the case (initial imaging study only). After power optimization, the Region of Interest (ROI) will be enlarged to collect data from the compartment of interest over 5 seconds and findings are averaged after processing. Both the fundamental data (B-mode data at 4 MHz) and the SHI data will be analyzed offline.

Exercise protocol: Patients will perform common exercise that causes symptoms is walking/running using a standardized exercise treadmill protocol: 3.7 mph against a 5° slope for 6 minutes or until symptom onset. If symptoms do not occur by 6 minutes of exercise, speed will be increased to a maximum of 5 mph and/or slope will be increased to 8° for an additional 6 minutes or until symptom onset. If the patient is still asymptomatic, he or she will exercise for another 4 minutes at 5 mph and an 8° slope or until symptom onset. Immediate post-exercise SWE and SHAPE will be performed using the same optimization parameters and protocol established for the pre-exercise portion of the study. Patients will be assigned a dummy code and de-identified SWE and SHI data will be stored for off line analysis.

The entire ultrasound portion of the study will last under 60 minutes and will be performed while the patient is under constant observation. The patient's vital signs will be monitored through the entire examination with frequent monitoring by the physician present. Active patient participation will conclude on completion of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* CECS as the primary diagnosis with no other more likely diagnoses.
* Age over 18.

Exclusion Criteria:

* Medial tibial stress syndrome or tibial stress fractures diagnosed on MRI.
* Recent trauma/surgery to the lower extremity
* Pregnant
* Stress fractures of the lower extremity
* Diabetic neuropathy
* Peripheral vascular disease
* Pressure ulcers or treatment for pressure ulcers
* Coronary artery disease
* Active pulmonary disease
* Allergy to any components of Definity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Accuracy in diagnosing | 2 years
  Evaluate the ability of SHAPE with microbubbles and SWE to accurately diagnose chronic exertional compartment syndrome (CECS) in percent using ROC analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request and approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code